CLINICAL TRIAL: NCT05675319
Title: Allogeneic Stem Cell Transplantation vs. Conventional Therapy as Salvage Therapy for Relapsed / Progressive Patients With Multiple Myeloma After First-line Therapy
Acronym: AlloRelapseMM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The reason for the end of recruitment is that the recruitment target could not be achieved despite all efforts and the G-BA (financing party) does not consider a continuation of the AlloRelapseMM study to be expedient.
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Gemeinsamer Bundesausschuss (G-BA) (Unknown); Staburo GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AlloRelapseMMStudy
Record Dates: First submitted 2022-11-06; First posted 2023-01-09 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: first relapse/progression after first-line therapy; allogeneic stem cell transplantation; salvage therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; elotuzumab; daratumumab; ixazomib; pomalidomide; isatuximab; selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (allo SCT) (Experimental): Allogeneic stem cell transplantation
  Interventions: Drug: Allogeneic Stem Cells
- Arm B (conventional therapy) (Active Comparator): Currently approved triple regimens for first relapse:
  * carfilzomib/lenalidomide/dexamethasone (KRD) or
  * elotuzumab/lenalidomide/dexamethasone (ERD) or
  * daratumumab/bortezomib/dexamethasone DVD) or
  * daratumumab/lenalidomide/dexamethasone (DRD) or
  * ixazomib/lenalidomide/dexamethasone (IRD) or
  * pomalidomide/bortezomib/dexamethasone (PVD) or
  * carfilzomib/daratumumab/dexamethasone (KDD) or
  * daratumumab/pomalidomide/dexamethasone (DPD) or
  * isatuximab/carfilzomib/dexamethasone (Isa-KD) or
  * selinexor/bortezomib/dexamethasone (SVD)
  Alternatively, autologous stem cell transplantation may also be performed, if sufficient stem cells are still cryopreserved.
  Interventions: Drug: carfilzomib/lenalidomide/dexamethasone (KRD); Drug: elotuzumab/lenalidomide/dexamethasone (ERD); Drug: daratumumab/bortezomib/dexamethasone (DVD); Drug: daratumumab/lenalidomide/dexamethasone (DRD); Drug: ixazomib/lenalidomide/dexamethasone (IRD); Drug: pomalidomide/bortezomib/dexamethasone (PVD); Drug: carfilzomib/daratumumab/dexamethasone (KDD); Drug: Autologous Stem Cells; Drug: daratumumab/pomalidomide/dexamethasone (DPD); Drug: isatuximab/carfilzomib/dexamethasone (Isa-KD); Drug: selinexor/bortezomib/dexamethasone (SVD)

INTERVENTIONS:
Drug: Allogeneic Stem Cells — Allogeneic Stem Cell Transplantation
  Arms: Arm A (allo SCT)
Drug: carfilzomib/lenalidomide/dexamethasone (KRD) — triple regimen for first relapse should be applied according to latest Summary of Product Characteristics (SmPC) version
  Arms: Arm B (conventional therapy)
Drug: elotuzumab/lenalidomide/dexamethasone (ERD) — triple regimen for first relapse should be applied according to latest SmPC version
  Arms: Arm B (conventional therapy)
Drug: daratumumab/bortezomib/dexamethasone (DVD) — triple regimen for first relapse should be applied according to latest SmPC version
  Arms: Arm B (conventional therapy)
Drug: daratumumab/lenalidomide/dexamethasone (DRD) — triple regimen for first relapse should be applied according to latest SmPC version
  Arms: Arm B (conventional therapy)
Drug: ixazomib/lenalidomide/dexamethasone (IRD) — triple regimen for first relapse should be applied according to latest SmPC version
  Arms: Arm B (conventional therapy)
Drug: pomalidomide/bortezomib/dexamethasone (PVD) — triple regimen for first relapse should be applied according to latest SmPC version
  Arms: Arm B (conventional therapy)
Drug: carfilzomib/daratumumab/dexamethasone (KDD) — triple regimen for first relapse should be applied according to latest SmPC version
  Arms: Arm B (conventional therapy)
Drug: Autologous Stem Cells — Autologous Stem Cell Transplantation
  Arms: Arm B (conventional therapy)
Drug: daratumumab/pomalidomide/dexamethasone (DPD) — triple regimen for first relapse should be applied according to latest SmPC version
  Arms: Arm B (conventional therapy)
Drug: isatuximab/carfilzomib/dexamethasone (Isa-KD) — triple regimen for first relapse should be applied according to latest SmPC version
  Arms: Arm B (conventional therapy)
Drug: selinexor/bortezomib/dexamethasone (SVD) — triple regimen for first relapse should be applied according to latest SmPC version
  Arms: Arm B (conventional therapy)

SUMMARY:
Allogeneic stem cell (allo SCT) transplantation for multiple myeloma is a potential curative treatment, but is associated with morbidity and treatment related mortality. Approved drug combinations or another autologous stem cell transplantation (auto-SCT) can be used for relapsed patients resulting in a median progression free survival up to 2-3 years.

In the current trial after first-line treatment relapsed or progressed myeloma patients with an HLA compatible donor will be randomized after 3 cycles of salvage therapy to allogeneic stem cell transplantation or to continuous conventional salvage therapy.

DETAILED DESCRIPTION:
The primary objective of the present clinical study aims to demonstrate the superiority of allogeneic stem cell transplantation (allo SCT) compared to conventional therapy for the difference in overall survival (OS) at 5 years in patients with multiple myeloma who have relapsed or progressed after first-line autologous hematopoietic stem cell therapy.

The secondary objectives are to show an improvement of progression free survival and relapse free survival after allo SCT compared to conventional therapy.

In addition, quality of life, toxicities, recurrence rates, non-relapse mortality (NRM), remission rates including minimal residual disease (MRD) and incidence of severe or life-threatening infection between the two arms are compared. Acute and chronic graft-versus-host disease (GvHD) after allo SCT are evaluated.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for study inclusion must meet criteria 1- 7 at registration and all of the following criteria before randomization:

1. Multiple Myeloma
2. Age 18 - 65 years
3. A signed informed consent form must be obtained before participation in the study
4. Age 66 - 70 years, if comorbidity index according to Sorror score = 0 and ECOG ≤ 1
5. 1st relapse/ progression according to IMWG criteria after first-line therapy (consisting of induction therapy followed by autologous transplantation once or twice and maintenance therapy), Additionally: meeting the need for treatment based on the SLiM-CRAB-criteria
6. Negative pregnancy test in female patients
7. Maximum of 1 cycle salvage therapy prior to study inclusion
8. Availability of a fully compatible stem cell donor (HLA-ident. Sibling or 10/10 MUD or 9/10 MMUD if mismatch affects DQB) after 3 cycles salvage therapy
9. CR/PR or SD according to IMWG-criteria after 3 cycles salvage therapy within the study

Exclusion Criteria:

Patients are excluded from the study if any one of criteria 1-6 are met at registration and if criterion 7 is met before randomization:

1. Non-sufficient organ function defined as:

   Bilirubin (in the absence of Meulengracht's disease), SGPT or SGOT ≥3 higher than normal values Cardiac ejection fraction ≤ 50% GFR < 30 ml/min DLCO < 35 % or continuous oxygen dependency
2. Active hepatitis B or C infection or uncontrolled HIV infection
3. Other, active malignant disease
4. Prior treatment with allogeneic stem cells
5. Participation in a clinical trial or taking an IMP within 30 days or five times the half-life of the IMP, whichever is longer, prior to registration
6. Positive serum pregnancy test at screening and before first treatment or breastfeeding
7. PD under salvage therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Overall survival at five years after randomization | at 5 years after randomization
  The present clinical study aims to demonstrate the superiority of allogeneic stem cell transplantation compared to conventional therapy for the difference in overall survival at 5 years in patients with multiple myeloma who have relapsed or progressed after first-line autologous hematopoietic stem cell therapy.

SECONDARY OUTCOMES:
Event-free survival at 1 year after randomization | from randomization to 1 year after randomization
  A secondary objective is to show an improvement of progress free survival and relapse free survival after allogeneic stem cell transplantation compared to conventional therapy.
  Events are defined as:
  * Progression or
  * Relapse or
  * Engraftment Failure or
  * Death of any cause
Event-free survival at 3 years after randomization | from randomization to 3 years after randomization
  A further secondary objective is to show an improvement of progress free survival and relapse free survival after allogeneic stem cell transplantation compared to conventional therapy.
  Events are defined as:
  * Progression or
  * Relapse or
  * Engraftment Failure or
  * Death of any cause
Event-free survival at 5 years after randomization | from randomization to 5 years after randomization
  A secondary objective is to show an improvement of progress free survival and relapse free survival after allogeneic stem cell transplantation compared to conventional therapy.
  Events are defined as:
  * Progression or
  * Relapse or
  * Engraftment Failure or
  * Death of any cause
Change from baseline in total EORTC score at 1 year after randomization | at visit Screening, at the end of cycle 3 (84 days, each cycle is 28 days) of salvage therapy, 6 months and 12 months after randomization
  The aim of the quality of life questionnaires (QLQ) is to provide a comparison between the two treatment arms. Quality of life according EORTC (European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) & Quality of Life Questionnaire - Multiple Myeloma Module (EORTC QLQ-MY20)) will be assessed in both groups..
  A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology/ sickness. Patients will be observed from baseline until database lock for final analysis and adjusted mean calculated at 1 year after randomization.
Change from baseline in total EORTC score at 3 years after randomization | at visit Screening, at the end of cycle 3 (84 days, each cycle is 28 days) of salvage therapy, 6 months, 1 year, 2 years and 3 years after randomization
  The aim of the quality of life questionnaires (QLQ) is to provide a comparison between the two treatment arms. Quality of life according EORTC (European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) & Quality of Life Questionnaire - Multiple Myeloma Module (EORTC QLQ-MY20)) will be assessed in both groups.
  A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology/ sickness. Patients will be observed from baseline until database lock for final analysis and adjusted mean calculated at 3 years after randomization.
Change from baseline in total EORTC score at 5 years after randomization | at visit Screening, at the end of cycle 3 (84 days, each cycle is 28 days) of salvage therapy, 6 months, 1, 2, 3, 4 and 5 years after randomization
  The aim of the quality of life questionnaires (QLQ) is to provide a comparison between the two treatment arms. Quality of life according EORTC (European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) & Quality of Life Questionnaire - Multiple Myeloma Module (EORTC QLQ-MY20)) will be assessed in both groups.
  A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology/ sickness. Patients will be observed from baseline until database lock for final analysis and adjusted mean calculated at 5 years after randomization.
Time to first occurrence of remission after randomization | at 30 days, 100 days, 6 months, 1 and 2 years after randomization
  Patients will be followed from randomization until database lock for final analysis and cumulative incidence of first remission (partial or complete), at 2 years after randomization, is reported.
Non-relapse mortality (NRM) at 1 year after randomization | from randomization to 1 year after randomization, an average of 1 year
  Patients will be observed from randomization until database lock for final analysis and cumulative incidence of death before any relapse at 1 year after randomization was reported.
Non-relapse mortality (NRM) at 3 years after randomization | from randomization to 3 years after randomization, an average of 3 years
  Patients will be observed from randomization until database lock for final analysis and cumulative incidence of death before any relapse at 3 years after randomization was reported.
Non-relapse mortality (NRM) at 5 years after randomization | from randomization to 5 years after randomization, an average of 5 years
  Patients will be observed from randomization until database lock for final analysis and cumulative incidence of death before any relapse at 5 years after randomization was reported.
Cumulative incidence of acute GvHD after allogeneic stem cell transplantation at 1 year after randomization | at 30 days, 100 days, 6 months and 1 year after randomization, an average of 1 year
  Patients will be observed from randomization until database lock for final analysis and cumulative incidence of any acute Graft-versus-Host Disease (GvHD, according to Przepiorka et al.) at 1 year after randomization is reported
Cumulative incidence of acute GvHD after allogeneic stem cell transplantation at 3 years after randomization | at 30 days, 100 days, 6 months, 1 year, 18 months and 2 years, 30 months and 3 years after randomization, an average of 3 years
  Patients will be observed from randomization until database lock for final analysis and cumulative incidence of any acute GvHD (according to Przepiorka et al.) at 3 years after randomization is reported
Cumulative incidence of acute GvHD after allogeneic stem cell transplantation at 5 years after randomization | at 30 days, 100 days, 6 months, 1 year, 18 months and 2 years, 30 months, 3, 4 and 5 years after randomization, an average of 5 years
  Patients will be observed from randomization until database lock for final analysis and cumulative incidence of any acute GvHD (according to Przepiorka et al.) at 5 years after randomization is repoted.
Cumulative incidence of chronic GvHD after allogeneic stem cell transplantation at 1 year after randomization | at 30 days, 100 days, 6 months and 1 year after randomization, an average of 1 year
  Patients will be observed from randomization until database lock for final analysis and cumulative incidence of any chronic GvHD (according to Jagasia et al.) at 1 year after randomization is reported.
Cumulative incidence of chronic GvHD after allogeneic stem cell transplantation at 3 years after randomization | at 30 days, 100 days, 6 months, 1 year, 18 months and 2 years, 30 months and 3 years after randomization, an average of 3 years
  Patients will be observed from randomization until database lock for final analysis and cumulative incidence of any chronic GvHD (according to Jagasia et al.) at 3 years after randomization is reported.
Cumulative incidence of chronic GvHD after allogeneic stem cell transplantation at 5 years after randomization | at 30 days, 100 days, 6 months, 1 year, 18 months and 2 years, 30 months, 3, 4 and 5 years after randomization, an average of 5 years
  Patients will be observed from randomization until database lock for final analysis and cumulative incidence of any chronic GvHD (according to Jagasia et al.) at 5 years after randomization is reported.
Time to first occurrence of infection reported as cumulative incidence of infection with CTCAE grade 3 - 5 at 1 year after randomization | from randomization to 1 year after randomization, an average of 1 year
  The severity and/or intensity of an adverse event will be graded based upon the patient's symptoms according to the current active version of National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE). Patients will be observed from randomization until database lock for final analysis and cumulative incidence of any infectious complication with CTCAE grade 3 - 5 at 1 year after randomization is reported.
Time to first occurrence of infection reported as cumulative incidence of infection with CTCAE grade 3 - 5 at 3 years after randomization | from randomization to 3 years after randomization, an average of 3 years
  The severity and/or intensity of an adverse event will be graded based upon the patient's symptoms according to the current active version of National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE). Patients will be observed from randomization until database lock for final analysis and cumulative incidence of any infectious complication with CTCAE grade 3 - 5 at 3 years after randomization is reported.
Time to first occurrence of infection reported as cumulative incidence of infection with CTCAE grade 3 - 5 at 5 years after randomization | from randomization to 5 years after randomization, an average of 5 years
  The severity and/or intensity of an adverse event will be graded based upon the patient's symptoms according to the current active version of National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE). Patients will be observed from randomization until database lock for final analysis and cumulative incidence of any infectious complication with CTCAE grade 3 - 5 at 5 years after randomization is reported.

OTHER OUTCOMES:
Event-free survival at 3 and 5 years after randomization | from randomization to 3 and 5 years after randomization
  Patients will be observed from randomization until database lock for interim analysis and the event-free survival (EFS) rate is calculated at 3 and 5 years after randomization.
  Events are defined as:
  * Progression or
  * Relapse or
  * Engraftment Failure or
  * Death of any cause
Change from baseline in total EORTC score (Summary Score) at 3 and 5 years after randomization | at visit Screening,at the end of cycle 3 (84 days, each cycle is 28 days) of salvage therapy, 6 months, 1, 2, 3, 4 and 5 years after randomization, an average at 3 and 5 years after randomization
  The aim of the quality of life questionnaires (QLQ) is to provide a comparison between the two treatment arms. Quality of life according EORTC (European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) & Quality of Life Questionnaire - Multiple Myeloma Module (EORTC QLQ-MY20)) will be assessed in both groups.
  A high score for a functional scale represents a high/ healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology/ sickness. Patients will be observed from baseline until database lock for interim analysis and adjusted mean is calculated at 3 and 5 years after randomization.
Non-relapse mortality at 1, 3 and 5 years after randomization | from randomization to 1, 3 and 5 years after randomization, an average of 1, 3 and 5 years
  Patients will be observed from randomization until database lock for interim analysis and cumulative incidence of death before any relapse at 1, 3 and 5 years after randomization is reported
Cumulative incidence of acute GvHD after allogeneic stem cell transplantation at 1, 3 and 5 years after randomization | at 30 days, 100 days, 6 months, 1 year, 18 months and 2 years, 30 months, 3, 4 and 5 years after randomization, an average of 1, 3 and 5 years
  Patients will be observed from randomization until database lock for interim analysis and cumulative incidence of any acute GvHD (according to Przepiorka et al.) at 1, 3 and 5 years after randomization is reported
Cumulative incidence of chronic GvHD after allogeneic stem cell transplantation at 1, 3 and 5 years after randomization | at 30 days, 100 days, 6 months, 1 year, 18 months and 2 years, 30 months, 3, 4 and 5 years after randomization, an average of 1, 3 and 5 years
  Patients will be observed from randomization until database lock for interim analysis and cumulative incidence of any chronic GvHD (according to Jagasia et al.) at 1, 3 and 5 years after randomization is reported
Time to first occurrence of Minimal Residual Disease (MRD) | at 30 days, 100 days, 6 months, 1 and 2 years after randomization, rate of occurence at 6 months, 1 and 2 years after randomization
  Patient observed from randomization until database lock for interim analysis and until database lock for final and rate of occurrence calculated at 6 months, 1 year and 2 years after randomization
Time to first occurrence of progression | from randomization to 1, 3, and 5 years after randomization
  Patients will be observed from randomization until database lock for interim analysis and rates at 3 and 5 years after randomization are calculated; and patients will be observed from randomization until database lock for final analysis and rates at 1, 3, and 5 years after randomization are calculated
Time to first recurrence of relapse | at 1, 3, and 5 years after randomization
  Patients will be followed from randomization to database lock for interim analysis and rates at 3 and 5 years after randomization are calculated; and patients will be followed from randomization to database lock for final analysis and rates at 1, 3, and 5 years after randomization are calculated.
Time to first occurrence of graft failure after stem cell transplatation | at day 30 after after randomization
  Patients are followed from randomization until database lock for interim analysis and rates at 3 and 5 years post-randomization are calculated; and patients are followed from randomization until database lock for final analysis and rates at 1, 3, and 5 years post-randomization are calculated. A graft failure is defined as no stable neutrophil count > 0.5 x 10^9/l at day 28 post-SCT.

CONTACTS AND LOCATIONS:
Overall Officials: Francis Ayuk, Prof. Dr. med., Principal Investigator — University Medical Center Hamburg-Eppendorf, Department of Stem Cell Transplantation
Locations (30):
- Germany (30):
  - University Hospital of Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg
  - Robert-Bosch Hospital Stuttgart, Stuttgart, Baden-Wurttemberg
  - University Hospital Tübingen, Tübingen, Baden-Wurttemberg
  - University Hospital of Ulm, Ulm, Baden-Wurttemberg
  - University Hospital Augsburg, Augsburg, Bavaria
  - University Hospital Munich ( LMU), München, Bavaria
  - University Hospital of the Technical University Munich rechts der Isar, München, Bavaria
  - Hospital North Nürnberg, Nuremberg, Bavaria
  - University Hospital Regensburg, Regensburg, Bavaria
  - University Hospital of Würzburg, Würzburg, Bavaria
  - Asklepios Hospital Hamburg St. Georg, Hamburg, Hamburg
  - University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg
  - University Hospital Frankfurt/ Main, Frankfurt am Main, Hesse
  - Philipps University Marburg, Marburg, Hesse
  - University Medical Center Göttingen, Göttingen, Lower Saxony
  - University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia
  - University Hospital Bonn, Bonn, North Rhine-Westphalia
  - University Hospital Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - University Hospital Essen, Essen, North Rhine-Westphalia
  - University Hospital Münster, Münster, North Rhine-Westphalia
  - Hospital Oldenburg (AöR), Oldenburg, Oldenburg
  - University Medical Center Mainz, Mainz, Rhineland-Palatinate
  - Hospital of Chemnitz gGmbH, Chemnitz, Saxony
  - University Hospital Carl Gustav Carus, Dresden, Saxony
  - University Hospital Halle (Saale), Halle, Saxony-Anhalt
  - University Hospital of Schleswig-Holstein (Campus Kiel), Kiel, Schleswig-Holstein
  - Charité - University of Medicine Berlin, Berlin, State of Berlin
  - Helios Hospital Berlin-Buch, Berlin, State of Berlin
  - University Hospital Jena, Jena, Thuringia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Glockner A, Schonland S, Einsele H, Kroger N. Rationale and design of the multicenter, national, randomized, open labeled phase III trial: allogeneic stem cell transplantation as a potential curative treatment for patients with relapsed or progressed multiple myeloma (AlloRelapseMM Study). BMC Cancer. 2025 Jan 27;25(1):147. doi: 10.1186/s12885-025-13503-7. PMID 39865222
- See also: Related Info — https://link.springer.com/article/10.1186/s12885-025-13503-7